CLINICAL TRIAL: NCT05531318
Title: Emotional Regulation in People With Co-occurring Posttraumatic Stress Disorder and Substance Use Disorder: A Qualitative Study of Individuals Receiving Community Substance Misuse Treatment
Brief Title: Emotional Regulation in People With Co-occurring Posttraumatic Stress Disorder and Substance Use Disorder
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Society for the Study of Addiction (Unknown)
Responsible Party: Sponsor
Other Study IDs: Bowen2022
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-03

CONDITIONS: Posttraumatic Stress Disorder; Substance Use Disorders; Emotional Regulation
Keywords: PTSD; Posttraumatic Stress Disorder; Substance Use Disorders; Trauma; Emotional regulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Emotional Regulation; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Qualitative Interview — Participants will be interviewed about their experiences of substance use, post-traumatic stress and the way they regulate their emotions.

SUMMARY:
The aim of this project is to look at emotional regulation in people with posttraumatic stress disorder (PTSD) and substance use disorder (SUD). This study will explore how people with PTSD-SUD regulate their emotions and how this might explain the relationship between these two disorders. In turn, this may inform effective treatment strategies for people with comorbid PTSD-SUD.

Emotional regulation refers to the way in which people process and respond to their emotions. PTSD and SUD commonly cooccur and this is associated with adverse outcomes including high rates of relapse, overdose, and suicide. We therefore need effective treatments to address this clinical concern. Evidence suggests emotional regulation might be important in the development and maintenance of PTSD and SUD and therefore it might be a useful target for treatment. However, most research in this area has been quantitative and has not considered how gender, social circumstances and trauma or substance type might affect the way people regulate their emotions. This study will recruit 40 adults with trauma histories and PTSD who are currently receiving treatment in a community drug and alcohol service for their substance use. Participants will be interviewed to explore how they regulate their emotions and how this relates to their social circumstances. This study will also explore whether gender, substance or trauma type affect the way people regulate their emotions. We hope this will help to improve treatment for people with PTSD and SUD.

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 18+

  * Receiving treatment from a community substance use service at the time of the study.
  * Experienced, witnessed or been confronted with at least one traumatic event (according to PTSD Diagnostic Scale for DSM-5) (PDS-5) (Foa, 2016).
  * Participant endorses at least 3 PTSD symptoms from criterion B-E, measured using the PDS-5.
  * Able to communicate and understand English sufficiently to engage in a qualitative interview.

Exclusion Criteria:

* • Staff recommend the individual should not take part in the study

  * The individual is unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample of approximately 40 people with posttraumatic stress disorder who are accessing substance use services in the community will be recruited and interviewed.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Qualitative interview accounts | November 2022 - October 2024
  Semi-structured interviews will be used

CONTACTS AND LOCATIONS:
Locations (1):
- National Addiction Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available to other researchers.

REFERENCES:
- [Background] Foa EB, McLean CP, Zang Y, Zhong J, Powers MB, Kauffman BY, Rauch S, Porter K, Knowles K. Psychometric properties of the Posttraumatic Diagnostic Scale for DSM-5 (PDS-5). Psychol Assess. 2016 Oct;28(10):1166-1171. doi: 10.1037/pas0000258. Epub 2015 Dec 21. PMID 26691504